CLINICAL TRIAL: NCT02692079
Title: The Effect of Titanium-Prepared Platelet-Rich Fibrin (T-PRF) Treatment on the Angiogenic Biomarkers in Gingival Crevicular Fluid (GCF) in Infrabony Defects of Patients With Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: The Effectiveness of Titanium-Prepared Platelet-Rich Fibrin on Angiogenic Biomarkers in Gingival Crevicular Fluid
Acronym: T-PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meltem Karsiyaka Hendek, Corresponding author, Clinical Research, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/18
Record Dates: First submitted 2016-02-18; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Periodontitis; Intrabony Periodontal Defect
Keywords: Angiogenesis; Bilateral infrabony defect; Flap surgery; Titanium-prepared, platelet-rich ﬁbrin
MeSH Terms: conditions — Chronic Periodontitis | interventions — Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-PRF+Allograft (Experimental): The defects were debrided and root planed with ultrasonic instrumentation and area-specific curets. All sites were washed with sterile salin solution and bleeding control was performed. Test group sites were treated with T-PRF+allograft
  Interventions: Procedure: T-PRF; Procedure: Allograft
- Allograft (Experimental): The defects were debrided and root planed with ultrasonic instrumentation and area-specific curets. All sites were washed with sterile salin solution and bleeding control was performed. Control group sites were treated with only allograft
  Interventions: Procedure: Allograft

INTERVENTIONS:
Procedure: T-PRF — Flap Surgery
  Arms: T-PRF+Allograft
Procedure: Allograft — Flap Surgery

SUMMARY:
This study investigates the effect of titanium-prepared platelet-rich fibrin (T-PRF) treatment on the angiogenic biomarkers in gingival crevicular fluid (GCF) in infrabony defects of patients with chronic periodontitis. In each patient, the infrabony defect of one side of arch was designated as control group (allograft), while the infrabony defect on the contralateral side of same arch was designated as test group (allograft+T-PRF).

DETAILED DESCRIPTION:
Platelets are the cells initiating the wound healing and also supporting it by secreting various growth factors actively. These growth factors released by platelets act the increase of connective tissue healing, bone regeneration and repair, fibroblast mitogenesis, wound angiogenesis and the activation of macrophages by stimulating cell proliferation signals.

Titanium-prepared, platelet-rich fibrin (T-PRF), is a new platelet concentrate, is formed in titanium tubes may be more efficient to activate platelets in comparison with glass tubes.The titanium tubes is utilized to refrain any inverse effects of glass tubes and also silica.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Chronic Periodontitis
* The presence of two or three-wall intrabony defects≥3 mm deep along with an interproximal probing depth ≥5 mm after non-surgical periodontal therapy

Exclusion Criteria:

* Systemic illnesses
* Any medications known to affect the outcomes of periodontal surgery
* Pregnancy and lactation

Ages: 26 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Platelet-derived growth factor-BB (ng/µl) , vascular endothelial growth factor-A (ng/µl), fibroblast growth factor-2 (ng/µl), anjiogenin (ng/µl), angiostatin (ng/µl) | Within the first 30 days after surgery

SECONDARY OUTCOMES:
The Volume of Gingival Crevicular Fluid (microliter) | Within the first 30 days after surgery

IPD SHARING:
Plan to Share IPD: No